CLINICAL TRIAL: NCT03604328
Title: An Open-label Phase I Study to Evaluate the Safety, Tolerability and Biodegradation Period of PolyActiva PA5108 Ocular Implant When Administered Intracamerally to the Anterior Chamber of the Eye
Brief Title: Safety and Tolerability of a Prostaglandin Ocular Implant for Treatment of Open Angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATA-CS101
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-03

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PA5108 (Experimental): PA5108 ocular implant (study eye) and topical prostaglandin analogue therapy (non-study eye)
  Interventions: Drug: PA5108

INTERVENTIONS:
Drug: PA5108 — single ocular implant, administered on day 1

SUMMARY:
A single centre, open label, study to assess the safety, tolerability and biodegradation of PA5108 ocular implant in adults who have Open Angle Glaucoma (Primary or Secondary).

DETAILED DESCRIPTION:
Participants who are currently managing their Open Angle Glaucoma with combination drop therapy will be recruited. Drop therapy will cease in the treatment eye and continue in the contralateral eye. The treated eye will receive via injection, a single PA5108 ocular implant. Participants will be monitored for safety and tolerability of the ocular implant until it completely biodegrades.

ELIGIBILITY:
Inclusion Criteria:

* Grade 3 or 4 open angle glaucoma (Shaffer-Etienne scale)
* Visual acuity in non-study eye same or better than study eye
* Currently taking topical ocular hypotensive medication including a prostaglandin analogue

Exclusion Criteria:

* Aphakic eyes
* Only one eye
* History of, or current uveitis, Cystoid Macular Edema (CME) or cornea edema
* Intraocular surgery or cornea/refractive surgery in study eye in past 6 months or anticipate need for eye surgery (including laser) in study eye during study period
* Current retinal detachment
* Uncontrolled infection in the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the occurrence of adverse events | 4 weeks

SECONDARY OUTCOMES:
Timeframe to complete implant biodegradation based on implant size and location | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Kerr, Principal Investigator — The Royal Victorian Eye & Ear Hospital
Locations (2):
- Australia (2):
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Melbourne Eye Specialists, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No